CLINICAL TRIAL: NCT00805779
Title: Pulsed Electromagnetic Stimulation for Treatment of Overactive Bladder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major protocol changes needeed
Sponsor: EMKinetics, Inc (Industry)
Responsible Party: Donna Deng, MD/Assistant Professor, UCSF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMK1208
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder; Overactive Urinary Bladder; Bladder, Overactive; Overactive Detrusor; Detrusor, Overactive; Overactive Detrusor Function; Detrusor Function, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MagPro R30 — Study treatments will be administered by a commercially available MagPro R30, with a cooled figure eight coil. The figure eight coil is placed directly over the posterior tibial nerve and the MagPro R30 will be activated. The coil will stimulate the posterior tibial nerve at 20 pulses per second for a 30 minute session.

SUMMARY:
To assess the initial safety and clinical feasibility of neuromodulation therapy in treating patients with documented overactive bladder. The specific aim is improved urinary frequency and urgency after 12 weeks of treatment

DETAILED DESCRIPTION:
Twenty to Forty patients with documented overactive bladder will receive 30 minutes of treatment one day a week for 12 weeks. Treatment will consist of stimulating the posterior tibial nerve in the area of the ankle with a pulsed electromagnetic field. Study treatments will be administered by a commercially available MagPro R30, with a cooled figure eight coil, and a surface electrode placed over the afferent pathway of the sacral nerve.

The specific aim is improved urinary frequency and urgency after 12 weeks of treatment.

Secondary goals.

* To estimate the extent to which the device will decrease the number of episodes of involuntary urine loss due to frequency/urgency in comparison to historical controls.
* To evaluate the potential of the device for improving patient quality of life as measured by a clinically validated scale, such as the Incontinence Quality of Life Instrument (I-QOL) or equivalent
* To periodically employ a micturition diary to record variables such as day/night urgency/frequency episodes, number of voids per day, severity of leaks, number of absorbent products used per day, etc.

ELIGIBILITY:
Inclusion Criteria:

* The patient is > 18 years old.
* The patient has ≥ 6 month history of documented overactive bladder.
* The patient has failed other conventional therapy (i.e.- Kegel exercises, biofeedback methodology, etc.).
* The patient is free of mechanical urethral obstruction as documented by cystoscopy or pressure flow criteria.
* The patient demonstrates an understanding of neuromodulation therapy, its benefits, and its potential risks.
* The patient is willing and able to keep accurate records of their voiding on the provided voiding diaries.
* The patient is willing and able to comply with the Study Protocol.
* The patient agrees to and is capable of answering a quality of life questionnaire.
* The patient has normal functioning of the upper urinary tract.
* The patient has an intact peripheral neurosensory system.
* If the patient is/was on pharmacologic treatment for urgency/frequency syndrome, a 10-day washout period prior to treatment must be completed.
* The patient has sufficient outlet resistance at the urinary sphincter (i.e.- the patient does not have intrinsic sphincter deficiency).

Exclusion Criteria:

* The patient is pregnant or intends to become pregnant during the course of the study. (Patients becoming pregnant during the course of the study will immediately be terminated from the study.) Warning: The effects of neuromodulation on a developing fetus are unknown
* The patient has an active urinary tract infection.
* The patient has abnormal cystoscopy, which is concerning for or indicative of malignancy.
* The patient has a urinary fistula.
* The patient has a bladder stone.
* The patient has had ankle injury or surgery which results inability to stimulate the tibial nerve or discomfort in using the foot cradle
* The patient has metal implant from surgery or a metallic foreign body in either leg below (distal to) the knee.
* The patient has cochlear implants.
* The patient has a hyperreflexic neurogenic bladder or urodynamically proven instability secondary to a known neurourologic cause (i.e.- stroke, Parkinson's, Multiple Sclerosis).
* The patient has had four or more urinary tract infections in the past year.
* The patient has a chronic disease or diminished mental capacity that, in the Principal Investigator's judgement, would impair their ability to successfully understand and comply with the protocol.
* The patient has a history of gross hematuria or glycosuria within the last year.
* The patient has chronic constipation (less than two (2) bowel movements per week).
* The patient has significant pathology that would compromise sphincter competency.
* The patient has uncontrolled diabetes.
* The patient has diagnosed peripheral neuropathy such as diabetes with peripheral nerve involvement.
* The patient has concomitant medical conditions that would limit the success of the procedure or confound study results, including but not limited to patients with nerve damage, pacemakers or implantable defibrillators.
* The patient is unable or unwilling to sign informed consent.
* The patient is on pharmacologic treatment that could affect bladder function.
* The patient has known moderate to severe ureteral reflux or hydronephrosis.
* The patient has severe urethral stricture(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Improved urinary frequency and urgency after 12 weeks of treatment. | 12 weeks

SECONDARY OUTCOMES:
To estimate the extent to which the device will decrease the number of episodes of involuntary urine loss due to frequency/urgency in comparison to historical controls | 12 weeks
To evaluate the potential of the device for improving patient quality of life as measured by a clinically validated scale, such as the Incontinence Quality of Life Instrument (I-QOL) or equivalent | 12 weeks
To periodically employ a micturition diary to record variables such as day/night urgency/frequency episodes, number of voids per day, severity of leaks, number of absorbent products used per day, etc | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donna Y Deng, MD, Principal Investigator — UCSF Department of Urology
Locations (1):
- UCSF Urology Faculty Practice, San Francisco, California, United States